CLINICAL TRIAL: NCT05944861
Title: Combination of Fluoroscopy and Ultrasonography Guidance in Sacroiliac Joint Injections: Effect on Procedure Time and Radiation Exposure
Brief Title: Combination of Fluoroscopy and Ultrasonography Guidance in Sacroiliac Joint Injections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Yasin Demir, Associate professor, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 35
Record Dates: First submitted 2023-03-15; First posted 2023-07-13 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2023-07

CONDITIONS: Sacroiliac Joint Somatic Dysfunction; Sacroiliac Joint Pain
Keywords: Sacroiliac joint pain; Sacroiliac joint injection; Ultrasonography guided injection; Flouroscopy guided injection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined ultrasonography and flouroscopy guided injeciton (Experimental): In 19 patients selected after randomization, the procedure will first be started with ultrasound and then continued with fluoroscopy.
  Interventions: Other: Combined ultrasonography and flouroscopy guided injeciton
- Flouroscopy guided injection (Active Comparator): In 19 patients selected after randomization, the procedure will be performed only through fluoroscopy.
  Interventions: Other: Flouroscopy guided injection

INTERVENTIONS:
Other: Combined ultrasonography and flouroscopy guided injeciton — In the ultrasound+fluoroscopy group, the sacroiliac injection will be started under ultrasound guidance. With the help of ultrasound, when sacral 2 foramen is seen the needle will be advanced to the entrance of the sacroiliac joint under real-time in-plane view. After considering intra-articular placement, fluoroscopy guidance will be initiated. An anteroposterior image will be taken to confirm whether contrast material is within the joint. If intra-articular placement is not achieved after contrast medium infiltration, needle reposition will be performed under fluoroscopy for correct needle placement. After the intraarticular contrast pattern is seen, 1 ml of 40 mg methylprednisolone + 1 ml of 1% lidocaine mixture will be injected.
  Arms: Combined ultrasonography and flouroscopy guided injeciton
Other: Flouroscopy guided injection — In the fluoroscopy group, the advancement of the needle into the sacroiliac joint will be performed by taking anteroposterior and lateral views. In the same way, the needle tip will be placed in the inferior of the sacroiliac joint, and contrast material distribution examination and injection of the drug will be performed as in the ultrasound + fluoroscopy group.
  Arms: Flouroscopy guided injection

SUMMARY:
The primary purpose of this study is to investigate the effect of the application of sacroiliac joint injection guided by combination of ultrasonography and fluoroscopy on the duration of the procedure and the amount of radiation exposed during the procedure, compared to the application of only fluoroscopy-guided technique. Secondary objectives are to evaluate the effectiveness of the treatment with both methods and to record the adverse events that may be encountered during the procedure.

DETAILED DESCRIPTION:
The study was designed as prospective, randomized, controlled trial. The patients who meet the eligibility requirements will be randomized into two groups in a 1:1 ratio to fluoroscopy and ultrasound+fluoroscopy. Processing time will be recorded during injection. "Fluoroscopy time" (sec) and "kerma-area product" (μGy) automatically measured by the fluoroscopy device will be used to evaluate the radiation exposure. Pre-procedural visual analogue scale (VAS) scores and Oswestry Disability Index (ODI) values were noted all the patients.

ELIGIBILITY:
Inclusion Criteria:

* Low back and/or gluteal pain and/or groin pain without radicular extension below the L4 level for more than 3 months
* Pain score greater than 3 according to NRS
* Unresponsiveness to conservative treatment (such as exercise, NSAID)
* At least 3 of the five sacroiliac provocation tests (FABER (Patrick), thigh thrust, Gaenslen, sacroiliac compression, and sacroiliac distraction tests) are positive

Exclusion Criteria:

Refusing to participate in the study

* Pregnancy
* Infective sacroiliitis
* Malignancy
* Osteoporosis
* Mechanical lumbosacral pathologies (spondylolisthesis, scoliosis, stenosis, etc.)
* Neurological finding in the lower extremity
* Pain spreading below the knee
* History of spinal surgery
* History of allergy to drugs to be injected (local anesthetic, contrast material, steroid allergy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Processing Time | during the intervention
  The processing time will be measured by the other researcher in the processing room with the help of a stopwatch. The stopwatch will be started when the needle touches the patient and will be stopped when the procedure is finished. It will be recorded in seconds

SECONDARY OUTCOMES:
Fluoroscopy Time | during the intervention
  The fluoroscopy time applied to the patient is automatically measured by the fluoroscopy device. This data will be saved
Kerma-area Product (μGy) | during the intervention
  The kerma area product will be measured to measure the radiation level to which the patient is exposed. This data is automatically measured by the fluoroscopy device.
Visual Analogue Scale | baseline, change from baseline VAS at 1 month after intervention
  Severity of pain was assessed using the standard 10 point VAS with 0 meant "no pain" at one end, and 10 meant "unbearable pain" at the other end
Oswestry Low Back Pain Disability Questionnaire | baseline, change from baseline VAS at 1 month after intervention
  The Oswestry disability index will be used to evaluate how much the patients' low back pain limits their activities in daily life. This index was first created in 1980 . The questionnaire consists of 10 sections, each assessing limitations in different daily activities and functions. Each section is scored from 0 to 5. A score of 0 indicates that there is no restriction while doing that activity, while a score of 5 represents the highest level of restriction in that activity. The maximum score is 50. As the total score increases, the disability level of the individual increases. In 2004, Turkish validity study was carried out by Yakut et al.

CONTACTS AND LOCATIONS:
Overall Officials: Serdar KESIKBURUN, MD, Principal Investigator — SBU,Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Locations (1):
- SBU,Gaziler Physical Medicine and Rehabilitation Education and Research Hospital, Ankara, Cankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No